CLINICAL TRIAL: NCT04436757
Title: Group Program IPS: Body-esteem and Self-esteem in a Psycho-social Rehabilitation Perspective
Brief Title: Self and Body-esteem in Socio-professional Rehabilitation
Acronym: IPS_FIRAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00777-32
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Bipolar Disorder; Personality Disorders; Anxiety Disorders; Depressive Disorder
Keywords: severe mental disorders; body-esteem; body-representation; self-esteem; socio-professional insertion
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Personality Disorders; Anxiety Disorders; Depressive Disorder; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, single-centre, comparative, interventional study, treated in open parallel groups, measuring the impact of "professional" body image intervention on improving body self-esteem in patients with severe mental health problems.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPS (Self-image and body-representation program) (Experimental): The IPS program (Self-image and body representation) was designed by Dr PLAZAT and coll. for specific use with patients with severe mental disorders suffering of low self- and body-esteem and aiming at " reinsert themselves" in the society.
  Interventions: Behavioral: IPS program : Self-image and body representation
- TAU (Active Comparator): Treatment As Usual : the usual care proposed by the health service (SUR/CL3R).
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: IPS program : Self-image and body representation — The IPS program consists in 13 sessions of 2 hours over a 13-weeks period.
  Sessions content is as follows :
  1. : Introduction
  2. : Sensory approach workshop
  3. : Self presentation and personal hygiene
  4. : Organisation of well-being, planning and pictograms
  5. : Becoming aware of my body, my envelope
  6. : Presentation and self-esteem (photolanguage)
  7. : Self-presentation in social interactions: Social codes
  8. : My ideas and desires for change
  9. : Places of well-being and clothing hygiene
  10. : Vocational insertion devices
  11. : Daring change : presence of a Socio-hairdresser
  12. : The awakening of color : presence of a Socio-aesthetician
  13. : Development of practice sheets and the network
  Arms: IPS (Self-image and body-representation program)
Behavioral: TAU — The treatment of the group TAU (Treatment As Usual) will consist of the usual care proposed by the health service. No additional session will be proposed.
  Arms: TAU

SUMMARY:
The body esteem influences the physical appearance, which can be a social brake. To enhance the socio-professional insertion of persons with severe mental disorders, the investigators developed a group program about self-presentation and body esteem. The study's objective is to understand the body esteem impact on socio-professional insertion, and how to improve that with a dedicated group program, for patients in a psychosocial rehabilitation center

DETAILED DESCRIPTION:
Our hypothesis is that a group program centered on the image and the presentation of the self, with the intervention of professionals of the image of the body, such as socio-hairdresser, socio-beautician, allows a better socio-professional inclusion, through an improvement in body self-esteem. Taking care of yourself will require different approaches such as advice on hygiene, becoming aware of your body, experimenting with beauty treatments and having the means to reproduce them at home. We will compare our IPS program (Image and Presentation of Self), with the usual management in the care center (TAU = "Treatment As Usual")

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65.
* Speaking French.
* Diagnosis of severe mental disorders (MSD) established according to the criteria of the DSM-V (Diagnostic and Statistical Manual of Mental Disorders) such as: Schizophrenia, Bipolar Disorders, Serious Personality Disorders, Severe Anxiety Disorders, Depressive Disorders; with a clinical stability of more than 3 months.
* Supported at SUR/CL3R with an application for socio-professional reintegration.
* Guardian agreement (for persons under guardianship);
* Information given to the curator (for persons under curatorship);
* Member of the social security scheme.

Exclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) or Eating Behaviour Disorder.
* Clinical status incompatible with group activity.
* Acute episode in progress.
* Refusal to participate.
* Simultaneous participation in a psycho-social rehabilitation program targeting image or self-esteem (general and/or body).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Appreciation of one's own appearance | baseline, one month, three months, nine months after the end of the treatment
  The main judgement criterion is the difference before/after the program for each of the two groups (IPS and TAU) of the weighted average at the "satisfaction with overall appearance" and "wish to change appearance" dimensions of the BES (Body-Esteem Scale), common dimensions for men and women. This difference will be compared between the 2 groups by a Student test (or a Wilcoxon-Mann-Whitney test in case of non normality).

SECONDARY OUTCOMES:
Appreciation of the Self-esteem measured by the Self-Esteem Rating Scale | baseline, one month, three months, nine months after the end of the treatment
  As for the primary outcome
Appreciation of the well-being measured by the Warwick-Edinburgh Well-Being Mental Scale | baseline, one month, three months, nine months after the end of the treatment
  As for the primary outcome
Appreciation of the satisfaction level measured by the Client's Assessment of Strengths, Interests and Goals Scale (CASIG ) | baseline, one month, three months, nine months after the end of the treatment
  As for the primary outcome
Appreciation of the satisfaction measured by the Satisfaction in the domains of life | baseline, one month, three months, nine months after the end of the treatment
  As for the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lucie-Orianne PLAZAT, M.D, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No